CLINICAL TRIAL: NCT04676607
Title: SHR7390 in the Treatment of Metastatic Hormone-Resistant Prostate Cancer That Failed Previous Docetaxel and New Endocrine Therapy
Brief Title: SHR7390 in Treating Patients With Metastatic Hormone-Resistant Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Hongqian Guo, Executive officer of Department of Urology, Drum Tower Hospital, Medical School of Nanjing University, Institute of Urology, Nanjing University, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: mCRPC-IIT-SHR7390
Record Dates: First submitted 2020-12-16; First posted 2020-12-21 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Metastatic Castration-resistant Prostate Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): SHR7390
  Interventions: Drug: SHR7390

INTERVENTIONS:
Drug: SHR7390 — SHR7390

SUMMARY:
This trial aims to prospectively assess the safety and efficiency of SHR7390 in metastatic castration-resistant prostate cancer

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-75 years，male
* ECOG PS：0-1
* Life expectancy of more than 6 months
* After surgery or drug castration, testosterone level was < 50 ng / dl. For subject receiving LHRH agonist / antagonist therapy (patients without orchiectomy), the treatment must start at least 4 weeks before the first day of cycle 1 and must be continued throughout the study
* Failure (radiological or PSA progression) or intolerance of at least one but not more than two taxanes based chemotherapy regimens and novel endocrine therapy (at least one of enzalutamide, apartamide, abitelone or shr3680). If docetaxel regimen used more than once, count as one regimen
* Disease progressed within 6 months prior to inclusion in the study. Disease progression defined as the occurrence of one or more of the following three items at the same time of castration：

  ① PSA progression，defined as at least twice increases in PSA level (interval time ≥ 1 week, and PSA level at screening should be ≥ 2ng / ml)

  ②Disease progression as defined in RECIST 1.1

  ③Bone disease progression defined by PCWG3，more than 2 new lesions in bone scan
* Metastatic lesions with radiologica evidence， measurable non-bone target lesions
* Adequate hepatic, renal, heart, and hematologic functions (no blood transfusion or hematopoietic growth factor treatment within 2 weeks before blood routine screening)：platelets>80×10^9/L，neutrophil>1.5×10^9/L, Hb≥90 g/L,total bilirubin≤1.5×limit of normal(ULN), ALT and AST ≤2.5×ULN（≤5×ULN with liver metastasis），blood urea nitrogen and creatinine≤1.5×ULN
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedure
* Willing to participate in this clinical trial, understand the research procedures and have signed informed consent

Exclusion Criteria:

* Prior treatment with MEK inhibitors，including trametinib
* Washout period from the end of any previous anti-tumor treatment (including radiotherapy, chemotherapy, surgery, molecular targeted therapy, immunotherapy, androgen receptor inhibitors, CYP-17 inhibitors, 5 α-reductase inhibitors, estrogen, progesterone drugs, etc) to the first administration of the study drug less than 1 week (bicalutamide elution period < 2 weeks)
* Plant drugs (e.g. Saw Palmetto) or steroids that may reduce PSA levels within 4 weeks, or planned to be used during the trial period (except for temporary steroid drugs for preventing or treating allergies)
* Plan to receive any other anti-tumor treatment during this trial
* Last drug administration from other clinical trials within 4 weeks
* Radiological confirmed tumor foci in the brain
* Severe bone injury caused by tumor bone metastasis judged by researchers, including severe bone pain with poor control, pathological fracture of important parts and spinal cord compression occurred or expected to occur in recent 6 months
* History of epilepsy, or the disease that can induce epilepsy within 12 months (including the history of transient ischemic attack, cerebral apoplexy (except for cerebral ischemic foci simply found by imaging examination), brain trauma with disturbance of consciousness and hospitalization）
* Hypotension (systolic blood pressure < 86mmhg) or uncontrollable hypertension (systolic blood pressure ≥ 150mmhg or diastolic blood pressure ≥ 100mmhg) within 30 days. The blood pressure results were the average value of three consecutive measurements with an interval of more than 2 minutes
* Active heart disease including severe/unstable angina pectoris, myocardial infarction, symptomatic congestive heart failure, and ventricular arrhythmias requiring drug treatment within 6 months
* Inability to swallow, chronic diarrhea and intestinal obstruction, or other factors affecting drug administration and absorption
* History of retinopathy confirmed by ophthalmic examination or neurosensory retinal detachment. Risk factors such as retinal vein thrombosis / occlusion (RVO), central serous retinopathy (CSR) or neovascular macular degeneration
* IOP > 21mmhg or diagnosed with glaucoma within 4 weeks
* Active HBV or HCV infection (HBV copies ≥ 10^4 copies / ml, HCV copies ≥ 10^3 copies/ml)
* History of immunodeficiency (including HIV positive, other acquired and congenital immunodeficiency diseases) or organ transplantation history
* Not willing to take effective contraceptive measures during the whole study period and within 6 months after the last administration
* Any accompanying diseases (such as poorly controlled hypertension, severe diabetes, thyroid disease and psychosis) that seriously endanger the safety of patients or affect the patients to complete the study

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-06-12 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 2 years
  The percentage of patients with measureable disease at baseline who achieved a complete or partial response in their soft tissue disease using the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria
AE | 2 years
  The type, frequency, severity, timing, seriousness, and relationship to study therapy

SECONDARY OUTCOMES:
PSA response rate | 2 years
  After the continuous therapy from randomisation to the end of the 12 weeks, the percentage of patients whose levels of PSA decreased by more than 50% compared with baseline
Time to prostate specific antigen (PSA) progression | 2 years
  Time from randomisation to the first time of PSA progression according to the criterion of PCGW3
Radiographic Progression Free Survival(rPFS) | 2 years
  Time from randomisation to radiologically confirmed progressive disease or death due to any cause
OS | 2 years
  Time from randomisation to death due to any cause
DoR | 2 years
  Time from radiologically confirmed reponse to radiologically confirmed progressive disease or death
Time to skeletal-related events | 2 years
  Time from randomisation to the first occurrence of a skeletal-related event. The skeletal-related event is defined as the occurrence of either pathological or clinical fracture, spinal cord compression, bone-related radiotherapy or surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hongqian Guo, Study Chair — Department of Urology, Drum Tower Hospital, Medical School of Nanjing University
Locations (1):
- The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China